CLINICAL TRIAL: NCT03792763
Title: Denosumab for High Risk SMM and SLiM CRAB Positive, Early Myeloma Patients- a Randomized, Placebo Controlled Phase II Trial "DEFENCE" (DEnosumab For the rEductioN of the Smoldering Myeloma transformatioN inCidence ratE)
Brief Title: Denosumab for High Risk SMM and SLiM CRAB Positive, Early Myeloma Patients
Acronym: DEFENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Amgen (Industry); Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGMT_MM-3
Record Dates: First submitted 2018-12-21; First posted 2019-01-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: early multiple myeloma; smoldering multiple myeloma; SLiM CRAB; denosumab; Austrian Study Group of Medical Tumour Therapy (AGMT); high risk smoldering myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: Placebo controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A, denosumab (Experimental): Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]
  Every 4 weeks (Q4W) for 6 months then every 3 months (Q3M) for a total of 3 years or until progression to active, symptomatic MM
  Calcilac 500 mg/400 I.E. (Calcium/Vitamin D3) Concomitant medication, oral, 1 chewable tablet / day
  Interventions: Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]
- Arm B, placebo (Placebo Comparator): Placebo 1.7 ml Subcutaneous Solution
  SC every 4 weeks (Q4W) for 6 months then every 3 months (Q3M) for a total of 3 years or until progression to active, symptomatic MM
  Calcilac 500 mg/400 I.E. (Calcium/Vitamin D3) Concomitant medication, oral, 1 chewable tablet / day
  Interventions: Drug: Placebo 1.7 ml Subcutaneous Solution

INTERVENTIONS:
Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA] — Administration every 4 weeks (Q4W) for 6 months then every 3 months (Q3M) for a total of 3 years or until progression to active, symptomatic MM
  Arms: Arm A, denosumab
Drug: Placebo 1.7 ml Subcutaneous Solution — Administration every 4 weeks (Q4W) for 6 months then every 3 months (Q3M) for a total of 3 years or until progression to active, symptomatic MM
  Arms: Arm B, placebo

SUMMARY:
This is a randomized, 2-arm phase II, placebo-controlled, multi-center study, where the investigators aim to evaluate whether the reported benefits of denosumab, delay of SRE and decrease in myeloma growth promotion, reduce the risk of progression of high-risk SMM and of early 'SLiM CRAB' myeloma into active, symptomatic CRAB positive myeloma or serological progression. In addition, tolerability of long-term treatment will be assessed.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether the transition of early Multiple Myeloma (High Risk Smouldering Multiple Myeloma SMM or "Ultra High Risk" SMM) or SLiM CRAB positive multiple myeloma to a symptomatic multiple myeloma (MM) can be reduced or delayed by the administration of denosumab.

With the exception of clinical studies, there are currently no standardized treatment options for SMM. Ultra-high risk SMM is already part of early active myeloma and is therefore in some cases treated according to a standard myeloma protocol (Revlimid-Dexamethasone, Velcade melphalan prednisone, melphalan prednisone thalidomide, or others). However, most practitioners recommend a wait-and-see strategy, since depending on the initial situation within two years only 58-95% of patients develop an 'active' MM and 5-42% of the patients had a stable disease and therefore do not necessarily have to be treated immediately.

Denosumab is a human monoclonal antibody (IgG2) which binds to RANKL with high affinity and specificity. RANKL (receptor activator of NF-κB Ligand) is a protein that is responsible for the formation, function and survival of osteoclasts (cell type responsible for bone resorption) Increased osteoclast activity, stimulated by RANKL, is a key mediator of the bone resorption in bone metastases and MM. Thus the activity of denosumab is resulting in a reduced number and function of osteoclasts and thus decreases the bone resorption and tumor-induced bone destruction.

After an initial phase of about 14 days (screening), the patients will be randomized 1:1 in one of the two study groups (arm A: denosumab or arm B: placebo). The study is double-blinded. The planned duration of therapy is 3 years. Patients receive denosumab or placebo every 4 weeks for 6 months, then every 3 months until a total of 3 years or progression.

After completion of the therapy, an observation and follow-up phase is carried out with patient visits every 3 months until the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to provide written informed consent in accordance with federal, local, and institutional guidelines
* Must meet criteria of high-risk smoldering MM or early "SLiM CRAB" MM based on the criteria described below:

  * High-risk SMM is defined here according to the revised Mayo Clinical criteria (2 out of 3 criteria must be fulfilled):

    * Bone marrow clonal plasma cells > 20%
    * Serum M protein > 2.0g/dL
    * Serum-free light chain ratio > 20, measured with "Binding site Kit"
  * Early 'SLiM CRAB' multiple myeloma

    * Patients must present with only one of the following features
    * Bone marrow clonal plasma cells ≥ 60%, or
    * Serum FLC ratio ≥ 100 (kappa-LC leading) or ≤ 0.01 (lambda-LC leading), measured with "Binding site Kit", or
    * >1 Focal bone lesion of ≥5mm (not associated with osteolysis, detected by PET-CT or whole-body low-dose CT (WBLDCT))
* Time from diagnosis of high-risk SMM or SLIM CRAB positive, early MM to study enrollment: <5 years

Exclusion Criteria:

* ECOG >3
* Active, symptomatic MM (fulfilling CRAB-criteria)
* Non-secretory MM, extramedullary plasmacytoma, plasma cell leukemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* MGUS
* Hypocalcemia (can be corrected by drug intervention before start of treatment)
* Second malignancy within the past 5 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer Gleason score ≤ 6 with stable prostate-specific antigen (PSA over 12 months)
  * Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins)
  * Treated medullary or papillary thyroid cancer
  * Similar condition with an expectation of > 95% five-year disease-free survival
* Active infection within the 14 days prior to randomization requiring systemic antibiotics and/or antiviral therapy
* Patients with known active or latent tuberculosis
* Known human immunodeficiency virus (HIV) seropositivity or active hepatitis C or hepatitis B infection (subjects with past hepatitis B virus [HBV] infection or resolved HBV infection defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test are eligible; subjects positive for hepatitis C virus [HCV] antibody are eligible only if polymerase chain reaction [PCR] is negative for HCV RNA.)
* Participation in another interventional study within the 28 days prior to randomization
* Any other clinically significant medical disease or social condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent, be compliant with study procedures, or provide accurate information.
* Prior administration of denosumab
* Prior exposure to any experimental or approved anti-myeloma agent
* Use of oral bisphosphonates with a cumulative exposure of more than 1 year (washout period for allowed bisphosphonate exposure 1 month)
* More than 1 previous dose of IV bisphosphonate or teriparatide administration (washout period for allowed bisphosphonate exposure 1 month)
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction
* Subject is pregnant or breastfeeding, or planning to become pregnant within 7 months after the end of treatment
* Female subject of childbearing potential is not willing to use, in combination with her partner, a highly effective and in addition an effective method of contraception during treatment and for 5 months after the end of treatment
* Known sensitivity to denosumab (including all components of the formulation) or any of the products to be administered during the study (eg, mammalian derived products, calcium, or vitamin D)
* Subject is receiving or is less than 30 days since ending other experimental devices or drugs (no marketing authorization for any indication).
* Subject will not be available for follow-up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Time to progression | 78 months (the first 6 cycles are 28 days, thereafter each cycle is 3 months for a maximum of 36 months)
  Time from randomization to transformation to symptomatic, active MM (defined as progression to active multiple myeloma according to IMWG diagnosis criteria 2014) or progression of disease according to IMWG response criteria 2016

SECONDARY OUTCOMES:
Percentage of patients transforming in 3 years | 36 months (the first 6 cycles are 28 days, thereafter each cycle is 3 months)
  Percentage of patients with high-risk SMM and early 'slim CRAB' positive MM transforming to CRAB positive multiple myeloma and/or developing serological progression (as defined by IMWG criteria 2016 for MM) within 3 years
Overall survival | 78 months (the first 6 cycles are 28 days, thereafter each cycle is 3 months for a maximum of 36 months)
  To determine the overall survival of patients receiving either denosumab or placebo
Time to first skeletal-related event | 78 months (baseline and every 6 months thereafter until progression or maximum of 3 years).
  To determine the time to first skeletal-related event for patients receiving either denosumab or placebo. • Imaging: low dose wbCT (details will be described in a separate guidance document) or PET-CT mandatory
Incidence of bone lesions as MM defining events | 78 months (baseline and every 6 months thereafter until progression or maximum of 3 years).
  To determine the incidence of bone lesions as MM defining events. • Imaging: low dose wbCT (details will be described in a separate guidance document) or PET-CT mandatory.
Time to first anti-myeloma treatment | 78 months (the first 6 cycles are 28 days, thereafter each cycle is 3 months for a maximum of 36 months)
  To determine the time to first anti-myeloma treatment for patients receiving either denosumab or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD, Study Director — Wilheminenspital
Locations (10):
- Austria (8):
  - IIIrd Medical Department, Private Medical University Hospital Salzburg, Salzburg, Salzburg
  - Medizinische Universitaet Graz, Univ.-Klinik f. Innere Medizin, Onkologie, Graz
  - Medizinische Universität Innsbruck Univ.-Klinik für Innere Medizin V Hämatologie und Onkologie, Innsbruck
  - LKH Hochsteiermark, Standort Leoben, Abteilung für Innere Medizin und Hämatologie und internistische Onkologie, Leoben
  - Kepler Universitaetsklinikum Klinik f. Interne 3, Med Campus III, Linz
  - BHS Linz: Interne I: Internistische Onkologie, Hämatologie und Gastroenterologie, Linz
  - Hanusch Krankenhaus der Österreichischen Gesundheitskasse, 3. Med. Abteilung, Vienna
  - Krankenhaus St. Vinzenz Zams, Innere Medizin, Internistische Onkologie und Hämatologie, Zams
- University Hospital Würzburg, Department of Internal Medicine 2, Würzburg, Germany
- Tel Aviv Sourasky Medical Center, Department of Hematology,, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakshman A, Rajkumar SV, Buadi FK, Binder M, Gertz MA, Lacy MQ, Dispenzieri A, Dingli D, Fonder AL, Hayman SR, Hobbs MA, Gonsalves WI, Hwa YL, Kapoor P, Leung N, Go RS, Lin Y, Kourelis TV, Warsame R, Lust JA, Russell SJ, Zeldenrust SR, Kyle RA, Kumar SK. Risk stratification of smoldering multiple myeloma incorporating revised IMWG diagnostic criteria. Blood Cancer J. 2018 Jun 12;8(6):59. doi: 10.1038/s41408-018-0077-4. PMID 29895887
- [Background] Mateos MV, Landgren O. MGUS and Smoldering Multiple Myeloma: Diagnosis and Epidemiology. Cancer Treat Res. 2016;169:3-12. doi: 10.1007/978-3-319-40320-5_1. PMID 27696254
- See also: Description sponsor — http://www.agmt.at